CLINICAL TRIAL: NCT05008497
Title: Validation in French of a Psychometric Tool for Measuring Health Literacy in the Field of Cancer
Brief Title: Cancer and Literacy in Health
Acronym: CaLiS
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A00421-40
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire

SUMMARY:
Validation in French of a psychometric tool for measuring health literacy in the field of cancer

DETAILED DESCRIPTION:
Single-centre, non-interventional questionnaire study

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older, having been informed of the research
* Followed or having been followed at the Hôpital privé des Peupliers for a cancer

Exclusion Criteria:

* Patient who has indicated his/her opposition to the use of his/her medical data
* Patient under legal protection, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients followed or having been followed for cancer at the Hôpital privé des Peupliers between May 2014 and December 2020
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Validation of a questionnaire | 6 months
  Development of the questionnaire: translation of the English version, testing of the French version in group work and then back-translation.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte NGO, MD PD, Principal Investigator — Hôpital Privé des Peupliers, Ramsay Santé
Locations (1):
- Hôpital Privé des Peupliers, Ramsay Santé, Paris, France

IPD SHARING:
Plan to Share IPD: No